CLINICAL TRIAL: NCT01004029
Title: A Phase 3B, Multi-Center, Randomized, Double-Blind Study of Hydroxyprogesterone Caproate (HPC) Injection, 250 mg/mL, Versus Vehicle for the Prevention of Preterm Birth in Women With a Previous Singleton Spontaneous Preterm Delivery
Brief Title: Confirmatory Study of 17P vs Vehicle for Prevention of Preterm Birth in Women w/ Previous Spontaneous Preterm Delivery
Acronym: PROLONG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AMAG Pharmaceuticals, Inc. (Industry)
Collaborators: ResearchPoint Global (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 17P-ES-003
Record Dates: First submitted 2009-10-27; First posted 2009-10-29 (Estimated); Results first posted 2021-01-28 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Preterm Birth
Keywords: 17P; 17-HPC; 17-OHPC; 17-hydroxyprogesterone caproate; progestogens; preterm birth; recurrent preterm birth; spontaneous preterm birth
MeSH Terms: conditions — Premature Birth | interventions — 17 alpha-Hydroxyprogesterone Caproate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vehicle (Placebo Comparator): Castor Oil
  Interventions: Drug: Vehicle
- Hydroxyprogesterone Caproate Injection (HPC), 250 mg/mL (Active Comparator): HPC 250 mg/mL in oil
  Interventions: Drug: Hydroxyprogesterone Caproate Injection (HPC), 250mg/mL

INTERVENTIONS:
Drug: Hydroxyprogesterone Caproate Injection (HPC), 250mg/mL — 1 mL intramuscular injection every week until 36 weeks, 6 days of gestation or delivery, whichever occurs first.
  Other Names: Makena; 17P
  Arms: Hydroxyprogesterone Caproate Injection (HPC), 250 mg/mL
Drug: Vehicle — Weekly intramuscular injections of 1 mL vehicle inert oil until 36 weeks, 6 days of gestation or delivery, whichever occurs first.
  Other Names: Placebo
  Arms: Vehicle

SUMMARY:
As part of the continuing effort to study the benefit and risks of 17P and preterm delivery, this study is designed as a multi-center, randomized, double-blind, vehicle-controlled clinical trial of 17P for the prevention of preterm birth prior to 35 weeks, 0 days of gestation in women with a singleton pregnancy, aged 18 years or older, with a previous singleton spontaneous preterm delivery. The study also includes a population pharmacokinetic (PK) substudy to assess the hydroxyprogesterone caproate (HPC) exposure-response relationship and the effect of body mass index (BMI) on the PK of 17P.

DETAILED DESCRIPTION:
One of the most significant risk factors for preterm birth is previous pregnancy history. Women who have had a prior preterm birth have a 2.5-fold greater risk than women with no prior history of preterm birth. Prophylactic methods for prevention of preterm birth, including tocolytic drugs, bed rest, and other interventions such as cerclage, have been shown in most studies to be ineffective. One of the preventive measures that has shown effectiveness in randomized trials is the use of progesterone agents.9,10 Progesterone has been shown to support gestation and to inhibit uterine activity.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet the following criteria to be enrolled in this study:

1. Age ≥ 18 years.
2. Singleton gestation.
3. Project gestational age 16 weeks 0 days of gestation or more and less than or equal to 20 weeks 6 days of gestation at the time of randomization, based on clinical information and evaluation of the first ultrasound.
4. Documented history of a previous singleton spontaneous preterm delivery. Spontaneous preterm birth is defined as delivery from 20 weeks 0 days to 36 weeks 6 days of gestation following spontaneous preterm labor or pPROM. Where possible, the gestational age of the previous preterm birth (referred to as the qualifying delivery) should be determined as described in "Gestational Age Determination". If the gestational age at delivery is obtained directly from the medical record and more than one gestational age appears, the latest will be used. As a validation of the gestational age of the previous delivery, if the infant weighed more than 3300 grams (the birth weight 90th percentile for 36 weeks gestational age), this will not qualify as preterm. The previous preterm delivery cannot be an antepartum stillbirth.

Exclusion Criteria:

1. Multifetal gestation.
2. Known major fetal anomaly or fetal demise. An ultrasound examination between 14 weeks 0 days through 20 weeks 3 days of gestation must be performed to rule out fetal anomalies.
3. Progesterone treatment in any form (i.e., vaginal, oral, intramuscular) during current pregnancy, other than micronized progesterone delivered orally or vaginally provided it is stopped at least 4 weeks prior to the first dose of study medication.
4. Heparin therapy during current pregnancy or history of thromboembolic disease.
5. Maternal medical/obstetrical complications including:

   * Current or planned cerclage
   * Hypertension requiring medication
   * Seizure disorder
6. Subjects with a uterine anomaly (uterine didelphys or bicornate uterus). However, subjects with uterine fibroids are eligible for the study.
7. Unwillingness to comply with and complete the study.
8. A 14 weeks 0 days through 20 weeks 3 days of gestation ultrasound cannot be arranged before randomization.
9. Participation in an antenatal study in which the clinical status or intervention may influence gestational age at delivery.
10. Participation in this trial in a previous pregnancy. Women who were screened in a previous pregnancy, but not randomized, do not have to be excluded.
11. Known hypersensitivity to hydroxyprogesterone caproate or its components.
12. Have any significant medical disorder that, in the opinion of the investigator, would be a contraindication to the use of the drug including those listed in section 5.3.2 of the investigational brochure. Other examples to consider include uncontrolled diabetes, known HIV infection or renal dysfunction.
13. Have any significant medical disorder that, in the opinion of the investigator, would preclude accurate evaluation of the subject's condition or outcome in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1740 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (103):
- United States (41):
  - Drug Research & Analysis Corporation, Montgomery, Alabama
  - Tucson Medical Center (Watching Over Mothers and Babies Foundation), Tucson, Arizona
  - Grossmont Center for Clinical Research, La Mesa, California
  - Naval Medical Center San Diego - Department of Obstetrics and Gynecology, San Diego, California
  - Womens Health Specialists, West Hills, California
  - Women's Associates, P.C., Colorado Springs, Colorado
  - Red Rocks OB/GYN - Physician's Research Options, LLC, Lakewood, Colorado
  - Visions Clinical Research, Boynton Beach, Florida
  - Palm Beach Obstetrics & Gynecology, PA (Altus Research), Lake Worth, Florida
  - Global OB/GYN Centers, Pembroke Pines, Florida
  - New Millennium Obstetrics & Gynecology, LLc, Riverdale, Georgia
  - Tripler Army Medical Center, Honolulu, Hawaii
  - The Women's Clinic, Boise, Idaho
  - Rosemark Women Care Specialists, Idaho Falls, Idaho
  - University of Louisville, Louisville, Kentucky
  - Women's Care Physicians/Obstetrical Specialists, PLLC, Louisville, Kentucky
  - Steven Z. Lenowitz, MD, LLC, Bel Air, Maryland
  - Female Pelvic Medicine and Urogynecology Institute of Michigan, Grand Rapids, Michigan
  - Saginaw Valley Medical Research Group, LLC, Saginaw, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Womack Army Medical Center, Fort Bragg, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Triad Research Partners, LLC, Winston-Salem, North Carolina
  - Mid Dakota clinicl, PC Center for Women, Bismarck, North Dakota
  - HWC Women's Research Center, Englewood, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - SC Clinical Research Center, LLC, Columbia, South Carolina
  - Greenville Hospital System University Medical Group, Greenville, South Carolina
  - Women's Physician's Group, MPLLC, Memphis, Tennessee
  - Practice Research Organization, Inc., Dallas, Texas
  - Carl R. Darnall Army Medical Center, Fort Hood, Texas
  - San Antonio Military Medical Center, Fort Sam Houston, Texas
  - Research Associates Rio Grande Valley, McAllen, Texas
  - Tanner Clinic, Layton, Utah
  - Mt. Timpanogos Women's Health Care, Pleasant Grove, Utah
  - Salt Lake Women's Center, P.C., Sandy City, Utah
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Madigan Army Medical Center, Tacoma, Washington
  - Wheaton Franciscan Healthcare - St. Joseph Campus, Milwaukee, Wisconsin
- Bulgaria (6):
  - MHAT "Blagoevgrad", Department of obstetrics and Gynecology, Blagoevgrad
  - Medical center "Teodora", LTD, Rousse
  - MHAT "Silistra", Obstetrics and Gynecology Department, Silistra
  - "Medical institute of Interior ministry", Sofia city PLC, Department of Gynecology, Sofia
  - Medical Centre "Avicena" Ltd, Sofia
  - SHAT " Sheinovo ",PLS, Maternity Clinic, Sofia
- Canada (6):
  - University of Calgary - Foothills Hospital, Calgary, Alberta
  - Lion's Gate Hospital (University of BC), North Vancouver, British Columbia
  - Glazier Medical Centre, Oshawa, Ontario
  - The Ottawa Hospital, General Campus, Ottawa, Ontario
  - Victory Reproductive Care, Windsor, Ontario
  - J. Leung Obstetrics and Gynaecology, Windsor, Ontario
- Czechia (6):
  - Fakultni nemocnice Olomouc, Olomouc, Olomoucký kraj
  - Fakultni nemocnice Brno, Brno, South Moravian
  - Nemocnice Ceske Budejovice, a.s. Gynekologicko-pordnicka klinika, České Budějovice
  - Fakultni nemocnice Hradec Kralove Porodnicka a gynekologicka klinika, Hradec Králové
  - Fakultni nemocnice Ostrava Porodnicko-gynekologicka klinika, Ostrava-Poruba
  - Fakultni nemocnice Pizen Gynekologicko-pordnicka klinika, Plzen-Lochotin
- Hungary (6):
  - Debreceni Egyetem Orvos es Egeszsegtudomanyi Centrum, Szuleszeti es Nogyogyaszati Klinika, Debrecen, Hajdú-Bihar
  - Fovarosi Onkormanyzat Egyesitett Szent Istvan es Szent Laszlo Korhaz-Rendelointezet, Szuleszet - Nogyogyaszat, Budapest
  - Petz Aladar Megyei Oktato Korhaz, Szuleszet-Nogyogyaszat, Győr
  - Bacs-Kiskun Megyei Onkormanyzat Korhaza, Svegedi Tudmanyegyetem Altalanos Orvostudomanyi kar Oktato Korhaza, Kecskemét
  - Josa Andras Oktato Korhaz Egeszsegugyi Szolgaltato Nonprofit Kft., Nyíregyháza
  - Szegedi Tudomanyegyetem, Szuleszeti es Nogyogyaszati Klinika, Szeged
- Italy (3):
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico S. Orsola-Malpighi, Bologna
  - Azienda Ospedaliera di Bolzano Ospedale Generale Regionale di Bolzano, Bolzano
  - Azienda Ospedaliera di Perugia - Ospedale Santa Maria dell a Misericordia, Perugia
- Russia (15):
  - Northern State Medical University, Arkhangelsk
  - Belgorod Regional Clinical Hospital of St.Ioasaf, Belgorod
  - State Educational Institution of Higher Professional Education "Kazan State Medical University of RosZdrav", Kazan'
  - Kemerovo State Medical Academy, Kemerovo
  - State Educational Institution of Higher Professional Education "Krasnoyarsk State University named After Prof. V.F. Voino-Yasenetsky of Ministry of Health Russia" Department of Perinatology, Obstetrics and Gynecology of Medical Faculty, Krasnoyarsk
  - State Educational Institution of Higher Professional Education "People's Friendship University of Russia" Department of Obstetrics and Gynecology with Course Perinatology, Moscow
  - Russian National Research Medical University named after N.I. Pirogov, Moscow
  - Municipal Healthcare Institution "Novosibirsk Municipal Perinatal Centre", Novosibirsk
  - Rostov Medical State University, Rostov-on-Don
  - State Educational Institution of Higher Professional Education "St. Petersburg l.l Mechnikov State Medical Academy of RosZdrav" Department of Obstetrics, Gynecology and Perinatology, Saint Petersburg
  - State Institution "D.O. Otto Scientific Institute for Obstetrics and Gynecology", Saint Petersburg
  - Almazov Federal Heart, Blood and Endocrinology Centre, Saint Petersburg
  - Regional Perinatal Center, Tomsk
  - State Healthcare Institution "Regional Maternity Hospital", Yaroslavl
  - Federal State Institution "Ural Research Institute of Maternity and Infancy Care of Rosmedtechnologies", Yekaterinburg
- Spain (8):
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Universitario Materno Infantil de Canarias, Las Palmas de Gran Canaria
  - Hospital Universitario La Paz, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Virgen Del Rocio, Seville
  - Hospital Universitario La Fe, Valencia
  - "Hospital Universitario Miguel Servet, Zaragoza
- Ukraine (12):
  - City Clinical Maternity Hospital #1, Chernivtsi
  - Donets'k Regional Centre of Mother and Child Care, Donets'k
  - Ivano-Frankivs'k Regional Prenatal Center, department of pregnant pathology, Ivano-Frankivsk
  - <<Institute of Pediatrics, Obstetrics and Gynecology of AMS Ukraine>> Department of Rehabilitation and Reproduktive function of Women, Kyiv
  - Polyclinic #1, Obolon district of Kyiv, maternity welfare department, Kyiv
  - Kyiv City Centre of Reproduction and perinatal medicine, obstetric department, Kyiv
  - SI "Institute of pediatrics, obstetrics and gynecology of AMS of Ukraine". Department of extragenital pathology and postnatal rehabilitation, Kyiv
  - Municipal Institution "Maternity Hospital #1", Odesa
  - Ternopil' Municipal Hospital # 2, Ternopil
  - Uzhgorod Municipal prenatal Centre, maternity welfare department #2, Uzhhorod
  - Clinical Maternity Hospital No 4, Zaporizhzhya
  - Department of Obstetrics and Gynecology of Zhaporizhzhya Medical Academy of Postgraduate Education on the Base of Healthcare Institution Maternity Hospital No 3, Zhaporizhzhya

REFERENCES:
- [Derived] Blackwell SC, Gyamfi-Bannerman C, Biggio JR Jr, Chauhan SP, Hughes BL, Louis JM, Manuck TA, Miller HS, Das AF, Saade GR, Nielsen P, Baker J, Yuzko OM, Reznichenko GI, Reznichenko NY, Pekarev O, Tatarova N, Gudeman J, Birch R, Jozwiakowski MJ, Duncan M, Williams L, Krop J. 17-OHPC to Prevent Recurrent Preterm Birth in Singleton Gestations (PROLONG Study): A Multicenter, International, Randomized Double-Blind Trial. Am J Perinatol. 2020 Jan;37(2):127-136. doi: 10.1055/s-0039-3400227. Epub 2019 Oct 25. PMID 31652479

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1740 subjects enrolled (signed the informed consent form), but only 1708 were randomized to each group (10 subjects did not return for Visit 2, 8 subjects did not meet all eligibility requirements, 8 subjects withdrew consent, and 6 subjects discontinued for other reasons).
Groups:
- 17P (Hydroxyprogesterone Caproate Injection): HPC 250 mg/mL in oil
  Hydroxyprogesterone Caproate Injection, 250mg/mL: 1 mL intramuscular injection every week until 36 weeks, 6 days of gestation or delivery, whichever occurs first.
Period: Overall Study
Arm/Group | Vehicle | 17P (Hydroxyprogesterone Caproate Injection)
Started (ITT Population - intent to treat) | 578 | 1130
Safety Population (Two subjects in the vehicle group were randomized to 17P but did not receive treatment with study medication.) | 578 | 1128
Completed (PP Population - per-protocol) | 530 | 1057
Not Completed | 48 | 73

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle | 17P (Hydroxyprogesterone Caproate Injection) | Total
Number analyzed (Participants) | 578 | 1130 | 1708
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.9 (5.22) | 30 (5.17) | 30.0 (5.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 578 | 1130 | 1708
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 101 | 155
  Not Hispanic or Latino | 524 | 1029 | 1553
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 22 | 23 | 45
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 41 | 73 | 114
  White | 504 | 1004 | 1508
  More than one race | 7 | 8 | 15
  Unknown or Not Reported | 4 | 18 | 22
Pre-pregnancy BMI (kg/m2), n [Mean (Standard Deviation); unit: kg/m^2] — Population: One participant did not have height recorded therefore BMI could not be calculated.
  kg/m^2
    number analyzed (Participants) | 577 | 1130 | 1707
    (all) | 24.7 (8.65) | 24.3 (7.05) | 24.5 (7.62)

OUTCOME MEASURES:

1. Primary Outcome: Preterm Birth <35 Weeks Gestation
Description: Determine if treatment with 17P reduces the rate of preterm birth < 35 weeks, 0 days of gestation in women with a previous singleton spontaneous preterm delivery.
Time Frame: Up to 35 weeks
Population: Number of ITT (intent to treat) subjects with non-missing delivery data or who were known to still be pregnant at 35 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | 17P (Hydroxyprogesterone Caproate Injection)
Number analyzed (Participants) | 574 | 1113
Participants | 66 | 122

2. Primary Outcome: Neonatal Composite Index (NCI)
Description: The composite index is defined as a liveborn neonate with any of the following occurring at any time during the birth hospitalization up through discharge from the NICU: neonatal death, grade 3 or 4 intraventricular hemorrhage, respiratory distress syndrome, bronchopulmonary dysplasia, necrotizing enterocolitis or proven sepsis.
Time Frame: Until 28 days of life or discharge from the neonatal intensive care unit (NICU), whichever occurred later.
Population: Liveborn Neonatal Population
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | 17P (Hydroxyprogesterone Caproate Injection)
Number analyzed (Participants) | 559 | 1093
Participants | 28 | 61

3. Secondary Outcome: Fetal/Early Infant Death
Description: Defined as spontaneous abortion/miscarriage (delivery from 16 weeks 0 days through 19 weeks 6 days of gestation) or neonatal death occurring in liveborns born at less than 24 weeks gestation or stillbirth (antepartum or intrapartum death from 20 weeks gestation through term), in the 17P group compared to the vehicle group
Time Frame: Delivery from 16 weeks 0 days through 19 weeks 6 days of gestation; or neonatal death occurring in liveborns born at less than 24 weeks gestation; or stillbirth (antepartum or intrapartum death) from 20 weeks gestation through term).
Population: Intent to Treat (ITT) Population - all randomized subjects regardless of whether they received study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | 17P (Hydroxyprogesterone Caproate Injection)
Number analyzed (Participants) | 578 | 1130
Participants | 11 | 19

4. Secondary Outcome: Preterm Birth Prior to 32 Weeks Gestation
Time Frame: Up to 32 weeks
Population: Intent to Treat (ITT) Population - all randomized subjects regardless of whether they received study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | 17P (Hydroxyprogesterone Caproate Injection)
Number analyzed (Participants) | 578 | 1130
Participants | 30 | 54

5. Secondary Outcome: Preterm Birth Prior to 37 Weeks Gestation
Time Frame: Up to 37 weeks
Population: Intent to Treat (ITT) Population - all randomized subjects regardless of whether they received study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | 17P (Hydroxyprogesterone Caproate Injection)
Number analyzed (Participants) | 578 | 1130
Participants | 125 | 257

6. Secondary Outcome: Stillbirths
Description: Defined as all stillbirths/fetal deaths/in utero fetal losses occurring from 20 weeks gestation until term.
Time Frame: 20 weeks gestation until term
Measure: Count of Participants; unit: Participants
Groups:
- Hydroxyprogesterone Caproate Injection, 250 mg/mL: HPC 250 mg/mL in oil
  Hydroxyprogesterone Caproate Injection, 250mg/mL: 1 mL intramuscular injection every week until 36 weeks, 6 days of gestation or delivery, whichever occurs first.
Arm/Group | Vehicle | Hydroxyprogesterone Caproate Injection, 250 mg/mL
Number analyzed (Participants) | 559 | 1093
Participants | 3 | 12

7. Secondary Outcome: Neonatal Deaths With ≥24 Weeks Gestational Age
Description: Neonatal death (from minutes after birth until 28 days of life) occurring in liveborns born at 24 weeks gestation or greater
Time Frame: Until 28 days of life or discharge from the NICU whichever occurred later.
Population: Liveborn Neonatal Population - all babies of randomized women who were liveborn and have morbidity data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | 17P (Hydroxyprogesterone Caproate Injection)
Number analyzed (Participants) | 558 | 1093
Participants | 2 | 3

ADVERSE EVENTS:
Time Frame: Randomized subjects were followed up to 35 ± 7 days after the last dose of study drug. Maternal and fetal deaths were reported until delivery if delivery occurred after 35 ± 7 days after last dose.
Description: Subjects reporting a particular adverse event (preferred term) or maternal pregnancy complication more than once are counted only once by preferred term and System Organ Class.
  All cause mortality used the ITT population. Serious and Other Adverse events used the Safety population.
Arm/Group | Vehicle | 17P (Hydroxyprogesterone Caproate Injection)
All-Cause Mortality (participants affected / at risk) | 0/578 | 0/1130
Serious Adverse Events (participants affected / at risk) | 18/578 | 34/1128
Other Adverse Events (participants affected / at risk) | 334/578 | 647/1128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle (N=578) | 17P (Hydroxyprogesterone Caproate Injection) (N=1128)
Cholestasis (Hepatobiliary disorders) | 3 | 0
Endometritis (Reproductive system and breast disorders) | 1 | 1
Escherichia sepsis (Infections and infestations) | 0 | 2
Migraine (Nervous system disorders) | 1 | 1
Placental insufficiency (Pregnancy, puerperium and perinatal conditions) | 1 | 4
Pneumonia (Infections and infestations) | 0 | 3
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 2 | 5
Pyelonephritis (Renal and urinary disorders) | 1 | 2
Wound infection (Infections and infestations) | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Pancreatitis relapsing (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Cholestasis of pregnancy (Hepatobiliary disorders) | 0 | 1
Amniotic cavity infection (Infections and infestations) | 0 | 1
Choriaoamnionitis (Infections and infestations) | 0 | 1
Clostridial infection (Infections and infestations) | 1 | 0
Endometritis (Infections and infestations) | 1 | 1
Endometritis decidual (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Mastitis postpartum (Infections and infestations) | 0 | 1
Pelvic abcess (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
bladder injury (Injury, poisoning and procedural complications) | 1 | 0
Incision site haematoma (Infections and infestations) | 1 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0
Biopsy chorionic villous abnormal (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Central nervous system inflammation (Nervous system disorders) | 0 | 1
Antepartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Confusion state (Psychiatric disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Scar (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Incision site haematoma (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle (N=578) | 17P (Hydroxyprogesterone Caproate Injection) (N=1128)
Anaemia (Blood and lymphatic system disorders) | 56 | 104
Anaemia of pregnancy (Blood and lymphatic system disorders) | 18 | 30
Abdominal pain (Gastrointestinal disorders) | 27 | 40
Abdominal pain lower (Gastrointestinal disorders) | 7 | 23
Constipation (Gastrointestinal disorders) | 17 | 38
Diarrhoea (Gastrointestinal disorders) | 13 | 23
Dyspepsia (Gastrointestinal disorders) | 25 | 37
Nausea (Gastrointestinal disorders) | 26 | 55
Vomiting (Gastrointestinal disorders) | 19 | 42
Injection site pain (General disorders) | 24 | 36
Injection site pruritus (General disorders) | 23 | 42
Oedema peripheral (General disorders) | 11 | 25
Nasopharyngitis (Infections and infestations) | 27 | 39
Urinary tract infection (Infections and infestations) | 23 | 44
Vaginal infection (Infections and infestations) | 21 | 41
Vaginitis bacterial (Infections and infestations) | 22 | 35
Vulvovaginal candidiasis (Infections and infestations) | 12 | 21
Gestational diabetes (Metabolism and nutrition disorders) | 21 | 33
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 50
Dizziness (Nervous system disorders) | 13 | 22
Headache (Nervous system disorders) | 28 | 68
Afterbirth pain (Pregnancy, puerperium and perinatal conditions) | 24 | 48
Cervical incompetence (Pregnancy, puerperium and perinatal conditions) | 16 | 34
Placental disorder (Pregnancy, puerperium and perinatal conditions) | 11 | 28
Insomnia (Psychiatric disorders) | 13 | 36
Shortened cervix (Reproductive system and breast disorders) | 15 | 18
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 17
Preeclampsia (Pregnancy, puerperium and perinatal conditions) | 22 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-04-06): https://cdn.clinicaltrials.gov/large-docs/29/NCT01004029/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-29): https://cdn.clinicaltrials.gov/large-docs/29/NCT01004029/SAP_001.pdf